CLINICAL TRIAL: NCT03424798
Title: Measuring Heart and Lung Function in Critical Care: A Feasibility Study to Assess the Use of a Novel Device to Monitor Cardiorespiratory Function in Mechanically Ventilated Patients in Critical Care.
Brief Title: Measuring Heart and Lung Function in Critical Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 212665
Record Dates: First submitted 2017-08-09; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Critical Illness; Mechanical Ventilation Complication; Haemodynamic Instability; Gas Exchange Impairment
Keywords: mechanical ventilation; lung function; cardiopulmonary monitoring
MeSH Terms: conditions — Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Inspiwave — patients are monitored with the Inspiwave device. A low dose inert tracer gas is added to the inspred air

SUMMARY:
This is a feasibility study of the use of a novel technique called 'Inspiwave' to measure heart and lung function in adult patients in critical care.

The preliminary work has already been undertaken in animal models and in healthy volunteers. The ultimate aim of this study is to develop a clinical tool for measuring (and therefore being able to make treatment changes based on) indices of heart and lung function in critical care patients. This study is the first assessment of the technique in this population, and whilst we know it works in patients undergoing general anaesthesia, we now need to assess whether Inspiwave can be used at all in critical care patients who may have much more physiological derangement. The purpose of this phase of the research is to determine whether it is feasible to use Inspiwave in critical care.

Inspiwave generates a sinusoidally modulated tracer gas signal in the inspired air. It also measures the resulting signal in the expired air. The unique handling of this signal by the patient can used be to derive key variables related to cardiopulmonary function such as lung volume, pulmonary blood flow, the deadspace (wasted ventilation) and the degree to which ventilation and blood flow are non-uniform. These are 'vital signs' in sick patients, yet are currently technically difficult to measure, particularly non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring mechanical ventilation in a critical care area

Exclusion Criteria:

* decision of participant not to be included
* consultee declaration not to be included
* Severely impaired gas exchange as declared by the managing clinician
* oxygen requirement exceeding 90% FIO2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -mechanically ventilated patients in a critical care area
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-21 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Production of any numerical values of effective lung volume and pulmonary blood flow | Sept 2020
  We wish to know whether the technique can be applied, and whether the signal to noise ratio allows computation of the variables of interest. It is yet unclear whether or not the device can operate in a critical care environment.

SECONDARY OUTCOMES:
Comparison of measurements of effective lung volume and pulmonary blood flow under changes in observed clinical condition. | Sept 2020
  To observe if changes in clinical condition can be detected by the device.
Signal:noise ratio of measured data. | Sept 2020
  If values for effective lung volume and pulmonary blood flow can be produced, are these with adequate signal:noise ratio to allow inverse modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Farmery, MD, Principal Investigator — heather.house@admin.ox.ac.uk
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No